CLINICAL TRIAL: NCT04341181
Title: ProTarget - A Danish Nationwide Clinical Trial on Targeted Cancer Treatment Based on Genomic Profiling
Acronym: ProTarget
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ulrik Lassen (Other)
Collaborators: Roche Pharma AG (Industry); Pfizer (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Ulrik Lassen, Professor, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ProTarget
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Tumors; Neoplasms; Neoplasia
MeSH Terms: conditions — Neoplasms | interventions — alectinib; atezolizumab; avelumab; Axitinib; Erlotinib Hydrochloride; Vemurafenib; cobimetinib; Trastuzumab; pertuzumab; Ado-Trastuzumab Emtansine; HhAntag691; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Alectinib (Experimental): Alectinib for patients with a molecular tumor profile that can potentially be targeted by Alectinib.
  Interventions: Drug: Alectinib
- Atezolizumab (Experimental): Atezolizumab for patients with a molecular tumor profile that can potentially be targeted by Atezolizumab.
  Interventions: Drug: Atezolizumab
- Avelumab (Experimental): Avelumab for patients with a molecular tumor profile that can potentially be targeted by Avelumab.
  Interventions: Drug: Avelumab
- Axitinib (Experimental): Axitinib for patients with a molecular tumor profile that can potentially be targeted by Axitinib.
  Interventions: Drug: Axitinib
- Erlotinib (Experimental): Erlotinib for patients with a molecular tumor profile that can potentially be targeted by Erlotinib.
  Interventions: Drug: Erlotinib
- Vemurafenib plus Cobimetinib (combination) (Experimental): Vemurafenib plus Cobimetinib (combination treatment) for patients with a molecular tumor profile that can potentially be targeted by Vemurafenib plus Cobimetinib.
  Interventions: Drug: Vemurafenib plus Cobimetinib (combination)
- Trastuzumab plus Pertuzumab (combination) (Experimental): Trastuzumab plus Pertuzumab (combination treatment) for patients with a molecular tumor profile that can potentially be targeted by Trastuzumab plus Pertuzumab.
  Interventions: Drug: Trastuzumab plus Pertuzumab (combination)
- Trastuzumab emtansin (Experimental): Trastuzumab emtansin for patients with a molecular tumor profile that can potentially be targeted by Trastuzumab emtansin.
  Interventions: Drug: Trastuzumab emtansine
- Vismodegib (Experimental): Vismodegib for patients with a molecular tumor profile that can potentially be targeted by Vismodegib.
  Interventions: Drug: Vismodegib
- Niraparib (Experimental): Niraparib for patients with a molecular tumor profile that can potentially be targeted by Niraparib.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Alectinib — Alectinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Alectinib might be expected based on their molecular tumor profile.
  Other Names: Alecensa
  Arms: Alectinib
Drug: Atezolizumab — Atezolizumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Atezolizumab might be expected based on their molecular tumor profile.
  Other Names: Tecentriq
  Arms: Atezolizumab
Drug: Avelumab — Avelumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Avelumab might be expected based on their molecular tumor profile.
  Other Names: Bavencio
  Arms: Avelumab
Drug: Axitinib — Axitinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Axitinib might be expected based on their molecular tumor profile.
  Other Names: Inlyta
  Arms: Axitinib
Drug: Erlotinib — Erlotinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Erlotinib might be expected based on their molecular tumor profile.
  Other Names: Tarceva
  Arms: Erlotinib
Drug: Vemurafenib plus Cobimetinib (combination) — Vemurafenib plus Cobimetinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Vemurafenib plus Cobimetinib might be expected based on their molecular tumor profile.
  Other Names: Zelboraf plus Cotellic (combination)
  Arms: Vemurafenib plus Cobimetinib (combination)
Drug: Trastuzumab plus Pertuzumab (combination) — Trastuzumab plus Pertuzumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Trastuzumab plus Pertuzumab might be expected based on their molecular tumor profile.
  Other Names: Herceptin plus Perjeta (combination)
  Arms: Trastuzumab plus Pertuzumab (combination)
Drug: Trastuzumab emtansine — Trastuzumab emtansine treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Trastuzumab emtansine might be expected based on their molecular tumor profile.
  Other Names: Kadcyla
  Arms: Trastuzumab emtansin
Drug: Vismodegib — Vismodegib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Vismodegib might be expected based on their molecular tumor profile.
  Other Names: Erivedge
  Arms: Vismodegib
Drug: Niraparib — Niraparib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Niraparib might be expected based on their molecular tumor profile.
  Other Names: Zejula
  Arms: Niraparib

SUMMARY:
The ProTarget study is a phase II, prospective, non-randomized clinical trial with the primary purpose of investigating the safety and efficacy of commercially available cancer drugs that target specific changes in cancer cell DNA to treat patients with advanced cancer. The primary endpoint is anti-tumor activity or stable disease documented after 16 weeks of experimental drug treatment. The drugs used in the trial have been approved by EMA/FDA for the treatment of certain cancers. Choice of drug is based on whether the patient's cancer cells contain precisely the DNA change (i) targeted by the EMA/FDA-approved drug or (ii) related to sensitivity to the EMA/FDA-approved drug. The trial drug is thus not approved by the EMA/FDA or in Denmark for the treatment of the patient's cancer - it is so-called "off-label use". The secondary purposes are:

* To detect side effects in patients treated with commercially available targeted cancer drugs.
* Performing biomarker analyzes, including (but not limited to) whole-genome analysis (WGS) on a fresh tumor tissue sample (biopsy) at baseline and progression.
* To investigate mechanisms of resistance using recurrent / serial fresh tumor biopsies for WGS and so-called liquid biopsies, which are blood samples in which the cancer cell DNA is analyzed.

The secondary endpoints include response duration, progression-free survival, and overall survival.

DETAILED DESCRIPTION:
The ProTarget study is a phase II, prospective, non-randomized clinical trial that aims to describe the safety and efficacy of commercially available, targeted anti-cancer drugs prescribed for treatment of patients with advanced cancer having a potentially actionable genomic variant revealed by a genomic test or immunohistochemistry test for protein overexpression performed in a laboratory accredited by the competent local regulatory authority. The study also aims to catalogue the choice of genomic test by clinical oncologists and learn about the utility of data collected through this study to develop hypotheses for future clinical trials. Eligible patients will have an advanced malignant disease with molecular aberrations for which standard treatment options are no longer available or feasible and acceptable performance status and organ function. A genomic test or immunohistochemistry test for protein overexpression must have been performed on a specimen of the tumor selected by the investigator in a laboratory accredited by the competent local regulatory authority and the test must identify at least one potentially actionable genomic variant as defined in the protocol. Genomic assays performed on cell-free DNA in plasma or other body fluids ("liquid biopsies") will also be acceptable if the genomic analysis is performed in a laboratory that meets the requirements described above. The investigator will select an appropriate drug from among those available in the protocol that targets the identified genomic variant and begin treatment once any drug-specific eligibility criteria are confirmed. If an eligible drug-variant match is not listed in the protocol, the physician may submit a proposal to treat with a drug available in the protocol, along with relevant clinical information and the genomic test results, to the study Molecular Tumor Board for review. The investigator may also choose to request options from the Molecular Tumor Board on treatment selection. The Molecular Tumor Board will return to the physician a list of potential treatment options. If the physician's choice of drug is among those available in the protocol and also one of the options provided by the Molecular Tumor Board, the protocol-specified treatment may be administered to the patient once any drug-specific eligibility criteria are confirmed. The investigator may not enroll a patient on a ProTarget study drug if it is not among the options listed in the protocol or provided by the Molecular Tumor Board. In this case, the non-ProTarget treatment and follow-up will be at the investigator's discretion. All patients who receive treatment with a drug available in the protocol will be followed for standard toxicity and efficacy outcomes including tumor response, progression-free and overall survival as well as duration of treatment and high grade or serious adverse events.

Study Objectives:

* To describe in different types of population the anti-tumor activity (efficacy) and toxicity (safety) of commercially available, targeted anti-cancer drugs used for treatment of patients with advanced disease with a genomic variant known (i) to be a target of an EMA-approved anti-cancer drug or (ii) to predict sensitivity to an EMA-approved anti-cancer drug.
* To record the site investigator determination treatment-related adverse events experienced by patients receiving treatment with commercially available, targeted anti-cancer drugs.
* To perform refined biomarker analyses, including (but not limited to) whole genome sequencing, on a fresh tumor biopsy specimen at baseline and at progression.
* To study mechanisms of resistance by the use of serial fresh tumor biopsies for WGS and liquid biopsies.

Study Population: Eligible patients will have an advanced malignant disease for which standard treatment options are no longer available or feasible and acceptable performance status and organ function. A genomic profiling test or immunohistochemistry test for protein expression or overexpression must have been performed on a specimen of the tumor in a laboratory accredited by the competent local regulatory authority. The results must identify at least one potentially actionable genomic variant that is targeted by a ProTarget Study drug, as defined in the protocol. Genomic assays performed on cell-free DNA in plasma ("liquid biopsies") will also be acceptable if the genomic analysis is performed in a laboratory that meets the requirements described above.

Intervention: Treatment with a commercially available, targeted anti-cancer drug matched to a genomic variant identified in a tumor biopsy specimen.

Study endpoints: Objective tumor response (complete response - CR or partial response- PR) or stable disease (SD) at 16 weeks or later after treatment initiation and safety are the primary study endpoints; progression-free survival, overall survival, duration of treatment on study and treatment-related high grade and serious adverse events will be collected.

Patients from Denmark, the Netherlands and the USA will be included in three similar though independent protocols (ProTarget, DRUP and TAPUR, respectively), allowing data-exchange and empowering of the trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (age≥ 18 years) with a histologically-proven locally advanced or metastatic malignant disease who is no longer benefitting from standard anti-cancer treatment or for whom, in the opinion of the investigator, no such treatment is available or indicated.
2. ECOG performance status 0-2
3. Patients must have acceptable organ function as defined below. However, as noted above, drug-specific inclusion/exclusion criteria specified in the appendix for each agent will take precedence for this and all inclusion criteria:

   1. Absolute neutrophil count ≥ 1500 µl
   2. Hemoglobin > 5.6 mmol/l
   3. Platelets > 75,000/µl
   4. Total bilirubin < 1.5 x institutional upper limit of normal (ULN)
   5. AST (SGOT) and ALT(SGPT) < 2.5 x institutional upper limit of normal (ULN) (or < 5 x ULN in patients with known hepatic metastases)
   6. Calculated or measured creatinine clearance ≥ 50 mL/min/1.73 m2.
4. Patients must have measurable or evaluable disease (per RECIST v1.1 for solid tumor), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or a subcutaneous or superficial lesion that can be measured with calipers by clinical exam. For lymph nodes, the short axis must be ≥15 mm. Patients who have assessable disease by physical or radiographic examination but do not meet these definitions of measurable disease are eligible and will be considered to have evaluable disease. Patient's whose disease cannot be objectively measured by physical or radiographic examination (e.g., elevated serum tumor marker only) are NOT eligible, with the exception of CA-125 for ovarian cancer and PSA for prostate cancer.
5. Results must be available from a genomic test or immunohistochemistry (IHC) test for protein expression performed in a laboratory accredited by the competent local regulatory authority. The genomic or IHC test used to qualify a patient for participation in ProTarget may have been performed on any specimen of the patient's tumor obtained at any point during the patient's care at the discretion of the patient's treating physician. Genomic assays performed on cell-free DNA in plasma ("liquid biopsies") will also be acceptable if the genomic analysis is performed in a laboratory accredited by the competent local regulatory authority.

   A new biopsy must be performed if possible, for central confirmation by WGS (the result may be awaited and is not required before first dosing).

   Note: Eligible genomic tests may include any of the following technologies: fluorescence in situ hybridization (FISH), polymerase chain reaction (PCR), comparative genomic hybridization (CGH), next generation sequencing (NGS), whole exome sequencing (WES). The test may have been performed on a fresh (frozen or in RNA-later) or paraffin-embedded specimen of the primary tumor or a metastatic deposit or on cell free DNA derived from plasma, as determined by the treating physician, and must reveal a potentially actionable genomic variant as defined in Section 5.0, or protein overexpression by IHC.
6. Ability to understand and the willingness to sign a written informed consent/assent document
7. Have a tumor genomic profile for which treatment with one of the approved targeted anti-cancer therapies included in this study has potential clinical benefit based on the criteria described in Section 7.0.
8. For orally administered drugs, the patient must be able to swallow and tolerate oral medication and must have no known malabsorption syndrome.
9. Because of the risks of drug treatment to the developing fetus, women of child-bearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) in combination with inhibition of ovulation (intrauterine device (IUD), intrauterine hormone-releasing system ( IUS), bilateral tubal occlusion, vasectomized partner or sexual abstinence) for the duration of study participation, and for four to 24 months following completion of study therapy (depending on SPC from individual drugs). Should a woman become pregnant or suspect she is pregnant while participating in this study or if she is the partner of a male participant in this study and becomes pregnant while he is participating in this study, she should inform her or her partner's treating physician immediately as well as her obstetrician. Female study patients who become pregnant must immediately discontinue treatment with any study therapy. Male patients should avoid impregnating a female partner. Male study patients, even if surgically sterilized, (i.e. post-vasectomy) must agree to one of the following: practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or completely abstain from sexual intercourse.

Exclusion Criteria:

1. Ongoing toxicity > CTCAE grade 2, other than peripheral neuropathy, related to anti-tumor treatment that was completed within 4 weeks prior to registration. Patients with ongoing peripheral neuropathy of ≥ CTCAE grade 3 will be excluded.
2. Previous treatment with the selected study drug for the same malignancy.
3. If the patient's tumor has a genomic variant known to confer resistance to an anti-cancer agent available in this study, the patient will not be eligible to receive that agent but will be eligible to receive other drugs available in this study if all inclusion and exclusion criteria are met for that drug.
4. Patient is receiving any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) except for medications that are prescribed for supportive care but may potentially have an anti-cancer effect (e.g., megestrol acetate, bisphosphonates) or ongoing castration-intent therapy for prostate cancer. These medications must have been started ≥ 1 month prior to enrollment on this study. Patients may be on warfarin, low molecular weight heparin or direct factor Xa inhibitors, unless such therapies are prohibited by drug-specific exclusion criteria.
5. Female patients who are pregnant or nursing. Male and female patients who refuse to practice highly effective contraception methods.
6. Patients with known progressive brain metastases determined by serial imaging or declining neurologic function in the opinion of the treating physician are not eligible. Patients with previously treated brain metastases are eligible, provided that the patient has not experienced a seizure or had a clinically significant change in neurological status within the 3 months prior to registration. All patients with previously treated brain metastases must be clinically stable for at least 1 month after completion of treatment and off steroid treatment for one month prior to study enrollment.

   Additional exclusion criteria specific for GBM patients:
   1. Patients who require anti-convulsant therapy must be taking non-enzyme inducing antiepileptic drugs (non-EIAED). EIAED are prohibited. Patients previously on EIAED must be switched to non-EIAED at least 2 weeks prior to randomization.
   2. No radiotherapy within the three months prior to the diagnosis of progression.
   3. No radiotherapy with a dose over 65 Gy, stereotactic radiosurgery or brachytherapy unless the recurrence is histologically proven.
7. Patients with preexisting cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias, or symptomatic congestive heart failure are not eligible.
8. Patients with left ventricular ejection fraction (LVEF) known to be < 40% are not eligible.
9. Patients with stroke (including TIA) or acute myocardial infarction within 4 months before the first dose of study treatment are not eligible
10. Patients with acute gastrointestinal bleeding within 1 month of start of treatment are not eligible.
11. Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements including, but not limited to: ongoing or active infection, significant uncontrolled hypertension, severe psychiatric illness situations, or anticipated or planned anti-cancer treatment or surgery.
12. Patients who do not meet drug-specific eligibility requirements for the drug selected by the investigator, are not eligible to receive that drug.
13. Patients whose disease is not measurable or assessable by radiographic imaging or physical examination (e.g., elevated serum tumor marker only) are not eligible.
14. Patients with known allergy/hypersensitivity to the study drug (active substance or to any of the excipients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 16 weeks
  Response according to RECIST

CONTACTS AND LOCATIONS:
Locations (7):
- Denmark (7):
  - Aalborg University Hospital, Aalborg, Aalborg
  - Aarhus University Hospital, Aarhus, Aarhus
  - Rigshospitalet, Copenhagen, Copenhagen
  - Herlev Hospital, Herlev, Herlev
  - Odense University Hospital, Odense, Odense
  - Zealand University Hospital, Roskilde, Roskilde
  - Vejle Sygehus, Vejle, Vejle

REFERENCES:
- [Derived] Kringelbach T, Hojgaard M, Rohrberg K, Spanggaard I, Laursen BE, Ladekarl M, Haslund CA, Harslof L, Belcaid L, Gehl J, Sondergaard L, Eefsen RL, Hansen KH, Kodahl AR, Jensen LH, Holt MI, Oellegaard TH, Yde CW, Ahlborn LB, Lassen U. ProTarget: a Danish Nationwide Clinical Trial on Targeted Cancer Treatment based on genomic profiling - a national, phase 2, prospective, multi-drug, non-randomized, open-label basket trial. BMC Cancer. 2023 Feb 22;23(1):182. doi: 10.1186/s12885-023-10632-9. PMID 36814246